CLINICAL TRIAL: NCT01773109
Title: Phase 2 Study of Etirinotecan Pegol (NKTR-102) in the Treatment of Patients With Metastatic and Recurrent Non-Small Cell Lung Cancer (NSCLC) After Failure of 2nd Line Treatment
Brief Title: Etirinotecan Pegol (NKTR-102) in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 18512
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Non Small Cell Lung Cancer; Recurrent Non Small Cell Lung Cancer
Keywords: Male/female subjects 18 years of age and older; metastatic or recurrent NSCLC; who failed 2nd line therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eligible patients will receive etirinotecan pegol at a dose of (Experimental): single-arm, open-label study is designed to investigate the efficacy and safety of etirinotecan pegol in patients with metastatic or recurrent NSCLC after failure of 2nd line therapy. Eligible patients will receive etirinotecan pegol at a dose of 145 mg/m2 iv every 3 weeks. One cycle will be defined as 3 weeks. Patients will be followed clinically every week for the first cycle with laboratory parameters (section 6.2.1) and physical exam. Response will be determined with RECIST version 1.1 after 2 cycles of therapy. Patients with Stable disease (SD), partial response (PR) or complete response (CR) will continue on additional therapy for up to six cycles. In the absence of disease progression in subjects completing six full cycles, further treatment beyond cycle #6 will be left to the discretion of the treating physician and his/her staff. Patients with progressive disease will be taken off study and will be followed for OS
  Interventions: Drug: Etirinotecan pegol (NKTR-102)

INTERVENTIONS:
Drug: Etirinotecan pegol (NKTR-102) — Eligible patients will receive etirinotecan pegol at a dose of 145 mg/m2 iv every 3 weeks. One cycle will be defined as 3 weeks. Treatment will be administered on an outpatient basis.
  Other Names: Etirinotecan Pegol (Topoisomerase I Inhibitor Polymer Conjugate) is a polyethylene glycol (PEG) conjugate of irinotecan.

SUMMARY:
This Phase 2 study is designed to characterize the objective response rate (defined as complete response (CR) and partial response (PR)) of Etirinotecan pegol administered to subjects with metastatic and recurrent NSCLC after failure of 2nd line therapy. Up to 37 eligible subjects will receive the investigational drug q3 weeks until they are no longer benefiting.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to characterize the objective response rate (defined as complete response (CR) and partial response (PR)) of Etirinotecan pegol (NKTR-102) administered to subjects with metastatic and recurrent NSCLC after failure of 2nd line therapy. Up to 37 eligible subjects will be enrolled at the University of Pennsylvania.

One cycle will be defined as 3 weeks. Patients will be followed clinically every week for the first cycle with laboratory parameters and physical exam. Response will be determined by RECIST version1.1 after 2 cycles of therapy. Patients with stable disease (SD), PR or CR will continue on treatment for up to six cycles. Those who are benefitting after six cycles will have the option of continuing on treatment. Patients with progressive disease will be taken off study and will be followed for OS data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or recurrent NSCLC. Primary or metastatic site may be used for histology.
* After failure of 2nd line treatment with up to two prior lines of therapy, one of which may be an oral TKI.
* Measurable disease (Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented incontrovertibly either radiographically or pathologically. For clinicians relying on biopsy documentation of recurrence, this must be obtained to confirm persistence at least 90 days following completion of radiation therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status is 0-1.
* Age at the time of study entry is ≥ 18 years.
* Adequate hematologic function as defined by an absolute neutrophil count (ANC) ≥ 1500/μL, hemoglobin ≥ 9.0 g/dL, and a platelet count ≥ 100,000/μL obtained within 2 weeks prior to enrollment.
* Adequate hepatic function as defined by a total bilirubin ≤ 1.5 mg/dL, and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 × the upper limit of normal ([ULN]), or ≤ 5 × the ULN in the presence of known liver metastases.
* Alkaline phosphatase (AP) ≤ 3 x the ULN or ≤ 5 × the ULN in the presence of known liver metastases
* Adequate renal function as defined by serum creatinine ≤ 1.5 × the institutional ULN. If creatinine is above the ULN, the patient's measured or calculated creatinine clearance (CrCl) must be ≥ 50 mL/min.
* Resolution of chemotherapy and radiation therapy related toxicities to NCI-CTCAE version 4.0 Grade 1 or lower severity, except for diarrhea (which must be Grade 0 without a supportive antidiarrheal medications) and alopecia (any grade).
* Women of childbearing potential and sexually active males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to enrollment and for the duration of study participation. Protections against pregnancy must be continued for at least 8 months after the last dose of study drug.
* Signed informed consent.

Exclusion Criteria:

* Untreated central nervous system metastases. Patients are eligible if they are clinically stable, off all steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, stereotactic radio surgery) ending at least 2 weeks prior to enrollment, or after surgical resection performed at least 2 weeks prior to enrollment.
* History of another "active" invasive primary cancer requiring ongoing treatment.
* Concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemo-embolization, targeted therapy, or an investigational agent.
* Patients who have had chemotherapy within 21 days (42 days for nitrosoureas or mitomycin C), radiotherapy within 14 days, biological therapy within 14 days, hormonal therapy within 7 days, and investigational therapy within 21 days prior to enrollment.
* Patients who have had any major surgery within 21 days prior to enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with chronic or acute GI disorders resulting in diarrhea of any severity grade; patients who are using chronic anti-diarrheal supportive care (more than 3 days/week) to control diarrhea in the 28 days prior to enrolment.
* Administration of the CYP3A4 inducers or inhibitors, as they may induce or inhibit irinotecan or SN38 metabolism within 14 days prior to cycle 1 and throughout study treatment. For a list of these agents, see: http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm
* Uncontrolled thrombotic or hemorrhagic disorder.
* Known human immunodeficiency virus (HIV) positivity.
* The patient, if female, is pregnant or lactating.
* Previous therapy with a topoisomerase I or II inhibitor.
* Known allergy to any of the treatment components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Etirinotecan Pegol: 145 mg/m2 will be administered as an IV infusion over a course of 90 minutes on Day 1 of a 21 day cycle
Period: Overall Study
Arm/Group | Etirinotecan Pegol
Started | 40
Completed | 37
Not Completed | 3
Not completed — Symptomatic Progression | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Etirinotecan Pegol: This Phase II, single-arm, open-label study is designed to investigate the efficacy and safety of etirinotecan pegol in patients with metastatic or recurrent NSCLC after failure of 2nd line therapy. Eligible patients will receive etirinotecan pegol at a dose of 145 mg/m2 iv every 3 weeks. One cycle will be defined as 3 weeks. Patients will be followed clinically every week for the first cycle with laboratory parameters and physical exam. Response will be determined with RECIST version 1.1 after 2 cycles of therapy. Patients with Stable disease (SD), partial response (PR) or complete response (CR) will continue on additional therapy for up to six cycles. In the absence of disease progression in subjects completing six full cycles, further treatment beyond cycle #6 will be left to the discretion of the treating physician and his/her staff. Patients with progressive disease will be taken off study and will be followed for overall survival.
Arm/Group | Etirinotecan Pegol
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 26
Age, Continuous [Median (Full Range); unit: years] | 66 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate
Description: The primary objective of this phase 2 trial is to estimate the objective response rate (Complete Response or Partial Response, as measured by RECIST version 1.1) for patients with metastatic or recurrent NSCLC being treated with etirinotecan pegol after failure of second-line therapy.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Etirinotecan Pegol
Number analyzed (Participants) | 37
Participants
  Partial Response | 2
  Stable Disease | 17
  Progressive Disease | 18

ADVERSE EVENTS:
Time Frame: 7 months
Description: As per CTCAE
Groups:
- Etirinotecan Pegol: Etirinotecan pegol (NKTR-102): 145mg/m2 intravenously every 3 weeks
Arm/Group | Etirinotecan Pegol
All-Cause Mortality (participants affected / at risk) | 37/40
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etirinotecan Pegol (N=40)
Treatment-related seconard maligancy (Nervous system disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic Event (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study failed to meet its prespecified response rate endpoint; thus, further studies with this agent are not planned at present.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes